CLINICAL TRIAL: NCT05369013
Title: Study and Follow-up of the Clinical Effectiveness and Comparative Safety of Biosimilar Teriparatide in the Management of Postmenopausal or Senile (ESECTO)
Brief Title: Study and Follow-up of the Clinical Effectiveness and Comparative Safety of Biosimilar Teriparatide in the Management of Postmenopausal or Senile.
Acronym: ESECTO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: STADA, Spain (Other)
Collaborators: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Instituto Palacios (Other); Complexo Hospitalario de Ourense (Other); Hospital Universitario Central de Asturias (Other); Parc Taulí Hospital Universitari (Other); Hospital Universitario Fundación Jiménez Díaz (Other); Hospital Universitario Infanta Leonor (Other); Hospital Universitario Virgen Macarena (Other); Hospital d´Igualada (Unknown); Alpha Bioresearch S.L. (Other)
Responsible Party: Sponsor
Other Study IDs: FHO-TER-2020-01
Record Dates: First submitted 2022-04-13; First posted 2022-05-11 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Risk fracture; Postmenopausical; Forsteo; Movymia
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Biosimilar Teriparatide
- B: Original Teriparatide

SUMMARY:
Non-interventional observational prospective follow-up study of cohorts of patients with Previous diagnosis of Osteoporosis with high risk of fractures, with/without previous fractures and treatment with bone formers (biosimilar or original Teriparatide), who meet all the inclusion criteria and exclusion, with prior information and signing of prior informed consent documents.

DETAILED DESCRIPTION:
Non-interventional observational prospective follow-up study of cohorts of patients with Previous diagnosis of Osteoporosis with high risk of fractures, with/without previous fractures and treatment with bone formers (biosimilar or original Teriparatide), who meet all the inclusion criteria and exclusion, with prior information and signing of prior informed consent documents.

Primary objective:

Verify the clinical effectiveness of Teriparatide Biosimilar under clinical practice conditions real. Compare this clinical effectiveness with original Teriparatide administered under similar conditions of actual clinical practice. Design: Observational cohort study, prospective, multicenter, nationwide. Study population: Patients with a previous diagnosis of Osteoporosis with a high risk of fractures,with/without previous fractures and in treatment with bone formers since before the start of the study. The patients will be distributed into 2 cohorts based on whether they are receiving similar Teriparatide (cohort A) or original Teriparatide (Cohort B).

ELIGIBILITY:
Inclusion Criteria:

* Signing the Informed Consent Men or women of legal age who have completed somatic growth.
* Previous diagnosis of densitometric osteoporosis in any location (densitometry with DEXA diagnosis within 6 months prior to start of treatment) or previous diagnosis of established osteoporosis (due to previous low-impact fracture, central or peripheral)
* Being in previous treatment with similar Teriparatide (cohort A) or with original Teriparatide (Cohort B).
* Be in possession of mental faculties to understand the therapeutic proposal, understand and follow the follow-up protocol and be able to sign the consent document informed.

Exclusion Criteria:

* The informed consent signature was not obtained.
* Patients who meet any of the contraindications for the use of teriparatide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with previous diagnosis of Osteoporosis with a high risk of fractures, with/without previous fractures and in treatment with bone formers since before the start of the study. The patients will be distributed into 2 cohorts based on whether they are receiving similar Teriparatide (cohort A) or original Teriparatide (Cohort B).
Sampling Method: Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-04-14 (Estimated)

PRIMARY OUTCOMES:
Effectiveness for patients treatment with original | 24 Months
  At the different moments of analysis (6, 12 and 24 months of treatment) in each of the treatment groups will be presented.
  The 95% confidence interval will be calculated for the mean percent change difference between groups. Likewise, the Student's t-test will be calculated for independent samples to assess statistical significance.
  To determine the fracture rate of any location during the study, the percentage of patients in each of the groups will be calculated descriptively. This proportion of patients will be compared between groups using Pearson's Chi-square test or Fisher's exact test, when applicable.
  The baseline-final change in biochemical markers of bone remodeling (BRM) between treatment groups will also be evaluated through the Student's t-test for independent samples if they meet the normality parameters or, failing that, its corresponding non-parametric test. (Mann-Whitney U test).
  .

SECONDARY OUTCOMES:
Confirm fracture rate in any localization while study is ongoing | 30 Months
  In order to determinate fracture rate from any localization, patient´s percentage from each group will be calculated in a descriptive way using: Bone fractures during treatment Falls.
Demographic and personal aspects related to the risk of osteoporosis | 24 Months
  age, sex, province of residence, year of diagnosis of OP.
Risk factor of osteoporosis | 30 Months
  As per previous patient´s medical records. Phisician will evaluated risk factor as per clinical practice. This information will be available at Clinical Records for each patients.
Previous clinical data | 24 Months
  Family history of interest as per clinical practice. This information will be available at Clinical Records for each patients.
Anthropometric clinical data | 24 Months
  weight and height will be combined to report BMI in kg/m^2
Osteoporosis diagnosis | 24 Months
  By BMD; BMD data in CL and hip, measured value in g/cm2 and T-Score value.
TBS | 24 Months
  TBS value
FRAX | 24 Months
  FRAX value of hip and major fracture.
Bone remodelling biomarkers | 24 Months
  Combined information described by: BGP (ng/ml), CTX (ng/ml), NTX (nmol/nmol creatine), P1NP (ng/ml), 25 OH vitamin D (ng/ml), intact PTH (pg/ml), TSH uUl/ml), Testosterone (ng/ml), Estradiol (pg/ml), Calcium (mg/dl), Phosphorus (mg/dl).This information will be collected in 194 patients who were recruited in this study. This information will be collected as per protocol during 30months. Physicians will evaluated this parameters as per clinical practice.
Hepatic profile | 24 Months
  Combined information described by: SGPT (U/L), SGOT (U/L), Gamma GT (U/L), FA (U/L), BT (mg/dl). This information will be collected in 194 patients who were recruited in this study. This information will be collected as per protocol during 30months. Physicians will evaluated this parameters as per clinical practice.
Previous bone fractures | 30 Months
  Number and type of previous fractures.
Previous treatment for osteoporosis | 24 Months
  Previous treatment of osteoporosis indicated as yes or no. This information will be available at Clinical Records for each patients.This information will be collected in 194 patients who were recruited in this study. This information will be collected as per protocol during 30months. Physicians will evaluated this parameters as per clinical practice.
Complementary previous treatment for osteoporosis | 24 Months
  Previous complementary treatment with Vitamin D and/or Calcium.
Security profile | 30 Months
  Number of secondary effects. Each secondary effects will be evaluted according to medical criterion.This information will be collected in 194 patients who were recruited in this study. This information will be collected as per protocol during 30months. Physicians will evaluated this parameters as per clinical practice. Day of start/end will be indicated.
Bone fractures during treatment | 24 Months
  Number of fractures during treatment.
Falls | 24 Months
  Number of falls during the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Palacios, Study Director — Instituto Palacios de la Salud de la Mujer. Presidente FHOEMO; Jose Luis Neyro, Study Director — Hospital Universitario Cruces. Embajador FHOEMO
Locations (10):
- Spain (10):
  - Hospital Parc Taulí, Barcelona
  - Hospital Universitario Igualada, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital de La Princesa, Madrid
  - Hospital Fundación Jimenez Diaz, Madrid
  - Hospital Infanta Leonor, Madrid
  - Instituto Palacio de Madrid, Madrid
  - Complejo Hospitalario Universitario de Orense, Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No